CLINICAL TRIAL: NCT00190398
Title: Endarterectomy Versus Angioplasty in Patients With Severe Symptomatic Carotid Stenosis
Brief Title: EVA3S: Endarterectomy Versus Angioplasty in Patients With Severe Symptomatic Carotid Stenosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Cecile jourdain, Department Clinical Research of developpement
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P990402
Record Dates: First submitted 2005-09-14; First posted 2005-09-19 (Estimated); Last update posted 2011-05-02 (Estimated); Status verified 2007-02

CONDITIONS: Transient Ischemic Attack; Carotid Stenosis; Atherosclerosis
Keywords: Prospective; Randomised; Open; Blinded End-point; PROBE Study; Ischemic stroke
MeSH Terms: conditions — Ischemic Attack, Transient; Carotid Stenosis; Atherosclerosis; Ischemic Stroke | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Carotid angioplasty and stenting with cerebral protection
  Interventions: Device: Carotid angioplasty and stenting with cerebral protection

INTERVENTIONS:
Device: Carotid angioplasty and stenting with cerebral protection — Carotid angioplasty and stenting with cerebral protection

SUMMARY:
The purpose of this study is to evaluate whether carotid angioplasty with stent (CAS) is as safe and effective as carotid surgery in regards to:

1. the risk of stroke and death within 30 days of the procedure;
2. the long-term risk of ipsilateral carotid territory stroke, in patients with recently symptomatic, severe carotid stenosis suitable for both CAS and carotid endarterectomy.

DETAILED DESCRIPTION:
Findings from two large randomized clinical trials - NASCET and ECST - have established endarterectomy as the standard treatment for severe symptomatic carotid artery stenosis. Compared to endarterectomy, stenting with or without cerebral protection has the advantage of avoiding general anesthesia and incision in the neck that could lead to nerve injury and wound complications. The costs may be less than those of surgery, mainly because of a shorter hospital stay. However, stenting also carries a risk of stroke and local complications. Unlike endarterectomy, which has known long-term benefits, stenting does not remove the atheromatous plaque, and the long-term efficacy of this technique needs also to be assessed. Several trials are in progress in Europe and the United States.

We established this trial to evaluate whether stenting is not inferior to endarterectomy concerning (a) the risk of stroke or death within 30 days of procedure and (b) the long-term risk of ipsilateral stroke, in patients with recently symptomatic, severe carotid stenosis.

ELIGIBILITY:
Inclusion Criteria:

* In brief, patients are eligible if they have experienced a carotid TIA or non disabling stroke within 4 months before randomisation and if they have an atherosclerotic stenosis of the region of the ipsilateral carotid bifurcation of 60% or more, as determined by the North American Symptomatic Carotid Endarterectomy Trial (NASCET) method, that investigators believe is suitable for both carotid endarterectomy and endovascular treatment. The degree of stenosis warranting treatment initially set at 70% or more was subsequently set at 60% or greater to reflect current generally accepted practice in the treatment of symptomatic carotid stenosis. The presence of a 60% or more ipsilateral carotid stenosis has to be confirmed by conventional digital subtraction angiography or the combination of carotid Duplex scanning and magnetic resonance angiography, provided the results of these non-invasive techniques are concordant.

Exclusion Criteria:

* Patients cannot be included if they have a disabling stroke (mRS >=3), a non atherosclerotic carotid disease, a severe intracranial carotid artery stenosis, contra-indications to heparin, ticlopidine or clopidogrel.
* There is no age limit.
* The presence of contralateral occlusion and/or the angiographic appearance of the stenotic lesion are not factors in treatment selection. The randomisation algorithm takes centre and degree of stenosis (more or less than 90% stenosis) into account. Patients must be treated as soon as possible after random assignment, in any case within 2 weeks of randomisation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2000-11; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Any stroke or death within 30 days of the procedure | during de study
  Any stroke or death within 30 days of the procedure

SECONDARY OUTCOMES:
Clinical: Myocardial infarction within 30 days of the procedure | during the study
  Clinical: Myocardial infarction within 30 days of the procedure
Other complications within 30 days of the procedure: cerebral (transient ischemic attack [TIA]) | during the study
  Other complications within 30 days of the procedure: cerebral (transient ischemic attack [TIA])
locoregional (e.g. cranial nerve palsy, complications at the site of puncture) | during the study
  locoregional (e.g. cranial nerve palsy, complications at the site of puncture)
General: Any disabling stroke or death within 30 days of the procedure plus disabling or fatal ipsilateral stroke during the follow-up period | during the study
  General: Any disabling stroke or death within 30 days of the procedure plus disabling or fatal ipsilateral stroke during the follow-up period
Any stroke or death within 30 days of the procedure plus any stroke (or any stroke or death) during the follow-up period | during the study
  Any stroke or death within 30 days of the procedure plus any stroke (or any stroke or death) during the follow-up period
TIA during the follow-up period | during the study
  TIA during the follow-up period
Functional status at the end of the study | during the study
  Functional status at the end of the study
Anatomical: Carotid restenosis (> 70% on carotid ultrasound) | during the study
  Anatomical: Carotid restenosis (> 70% on carotid ultrasound)
Integrity of the stent 2 years after the procedure (on cervical radiogram) | during the study
  Integrity of the stent 2 years after the procedure (on cervical radiogram)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis MAS, Pr, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Sainte-Anne Hospital: Department of Neurology, Paris, Île-de-France Region, France

REFERENCES:
- [Result] Mas JL, Chatellier G, Beyssen B, Branchereau A, Moulin T, Becquemin JP, Larrue V, Lievre M, Leys D, Bonneville JF, Watelet J, Pruvo JP, Albucher JF, Viguier A, Piquet P, Garnier P, Viader F, Touze E, Giroud M, Hosseini H, Pillet JC, Favrole P, Neau JP, Ducrocq X; EVA-3S Investigators. Endarterectomy versus stenting in patients with symptomatic severe carotid stenosis. N Engl J Med. 2006 Oct 19;355(16):1660-71. doi: 10.1056/NEJMoa061752. PMID 17050890
- [Derived] Howard VJ, Algra A, Howard G, Bonati LH, de Borst GJ, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Greving JP, Halliday A, Hendrikse J, Jansen O, Brown MM, Mas JL, Ringleb PA, Brott TG; Carotid Stenosis Trialists' Collaboration. Absence of Consistent Sex Differences in Outcomes From Symptomatic Carotid Endarterectomy and Stenting Randomized Trials. Stroke. 2021 Jan;52(2):416-423. doi: 10.1161/STROKEAHA.120.030184. Epub 2021 Jan 25. PMID 33493046
- [Derived] Muller MD, von Felten S, Algra A, Becquemin JP, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Halliday A, Hendrikse J, Howard G, Gregson J, Jansen O, Brown MM, Mas JL, Brott TG, Ringleb PA, Bonati LH. Secular Trends in Procedural Stroke or Death Risks of Stenting Versus Endarterectomy for Symptomatic Carotid Stenosis. Circ Cardiovasc Interv. 2019 Aug;12(8):e007870. doi: 10.1161/CIRCINTERVENTIONS.119.007870. Epub 2019 Aug 5. PMID 31378071
- [Derived] Muller MD, von Felten S, Algra A, Becquemin JP, Brown M, Bulbulia R, Calvet D, Eckstein HH, Fraedrich G, Halliday A, Hendrikse J, Gregson J, Howard G, Jansen O, Mas JL, Brott TG, Ringleb PA, Bonati LH; Carotid Stenosis Trialists' Collaboration. Immediate and Delayed Procedural Stroke or Death in Stenting Versus Endarterectomy for Symptomatic Carotid Stenosis. Stroke. 2018 Nov;49(11):2715-2722. doi: 10.1161/STROKEAHA.118.020684. PMID 30355202
- [Derived] Rantner B, Kollerits B, Roubin GS, Ringleb PA, Jansen O, Howard G, Hendrikse J, Halliday A, Gregson J, Eckstein HH, Calvet D, Bulbulia R, Bonati LH, Becquemin JP, Algra A, Brown MM, Mas JL, Brott TG, Fraedrich G; Carotid Stenosis Trialists' Collaboration. Early Endarterectomy Carries a Lower Procedural Risk Than Early Stenting in Patients With Symptomatic Stenosis of the Internal Carotid Artery: Results From 4 Randomized Controlled Trials. Stroke. 2017 Jun;48(6):1580-1587. doi: 10.1161/STROKEAHA.116.016233. Epub 2017 Apr 28. PMID 28455318
- [Derived] Mas JL, Arquizan C, Calvet D, Viguier A, Albucher JF, Piquet P, Garnier P, Viader F, Giroud M, Hosseini H, Hinzelin G, Favrole P, Henon H, Neau JP, Ducrocq X, Padovani R, Milandre L, Rouanet F, Wolff V, Saudeau D, Mahagne MH, Sablot D, Amarenco P, Larrue V, Beyssen B, Leys D, Moulin T, Lievre M, Chatellier G; EVA-3S Investigators. Long-term follow-up study of endarterectomy versus angioplasty in patients with symptomatic severe carotid stenosis trial. Stroke. 2014 Sep;45(9):2750-6. doi: 10.1161/STROKEAHA.114.005671. Epub 2014 Jul 31. PMID 25082808
- [Derived] Rantner B, Goebel G, Bonati LH, Ringleb PA, Mas JL, Fraedrich G; Carotid Stenting Trialists' Collaboration. The risk of carotid artery stenting compared with carotid endarterectomy is greatest in patients treated within 7 days of symptoms. J Vasc Surg. 2013 Mar;57(3):619-626.e2; discussion 625-6. doi: 10.1016/j.jvs.2012.08.107. Epub 2012 Dec 11. PMID 23237679
- [Derived] Mas JL, Trinquart L, Leys D, Albucher JF, Rousseau H, Viguier A, Bossavy JP, Denis B, Piquet P, Garnier P, Viader F, Touze E, Julia P, Giroud M, Krause D, Hosseini H, Becquemin JP, Hinzelin G, Houdart E, Henon H, Neau JP, Bracard S, Onnient Y, Padovani R, Chatellier G; EVA-3S investigators. Endarterectomy Versus Angioplasty in Patients with Symptomatic Severe Carotid Stenosis (EVA-3S) trial: results up to 4 years from a randomised, multicentre trial. Lancet Neurol. 2008 Oct;7(10):885-92. doi: 10.1016/S1474-4422(08)70195-9. Epub 2008 Sep 5. PMID 18774745